CLINICAL TRIAL: NCT02094482
Title: Prospective Evaluation of a New Palatal Implant for Treatment of Snoring and Obstructive Sleep Apnea (OSAS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medartis AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P08138.1
Record Dates: First submitted 2014-03-20; First posted 2014-03-21 (Estimated); Last update posted 2021-09-13 (Actual); Status verified 2021-09

CONDITIONS: Reduction of Initial AHI; Reduction of Initial Snoaring Index

ARMS (1):
- OSAS Palatal Implant (Other): The IMD is a resilient palatal implant which is introduced through a stab incision into the palate. Two implants are placed underneath the rostral part of the palatal bone and continue into the upper part of the soft palate .
  Interventions: Device: The IMD is a resilient palatal implant which is introduced through a stab incision into the palate.

INTERVENTIONS:
Device: The IMD is a resilient palatal implant which is introduced through a stab incision into the palate. — The IMD is a resilient palatal implant which is introduced through a stab incision into the palate. Two implants are placed underneath the rostral part of the palatal bone and continue into the upper part of the soft palate

SUMMARY:
Prospective Evaluation of a New Palatal Implant for Treatment of Snoring and Obstructive Sleep Apnea (OSAS)

DETAILED DESCRIPTION:
The new OSAS Implant is intended for use in the palate (hard and soft palate/ see picture above) in order to stiffen and stabilize the soft palate, which may reduce the severity of airway obstructions and of snoring in patients suffering from OSA (Obstructive Sleep Apnea). Indications for use of the System include: symptomatic, habitual, social snoring due to palatal flutter or upper airway obstruction primarily caused by the retropalatal obstruction. The System is labeled for use by physicians only.

The primary endpoint is the Apnea-Hypopnea-Index (AHI) in the 90 days follow-up.

Study hypothesis: Reduction of initial AHI ≥20%

ELIGIBILITY:
Inclusion Criteria:

Study patients must meet all of the following inclusion criteria:

* Socially disturbing snoring with/without obstructive sleep apnea syndrome
* Predominantly retropalatal obstructions established by ApneaGraph ≥60%, sleep nasendoscopy or successful application of the Velumount palatal device
* Findings for predominantly retropalatal obstructions in ENT-examination:
* No tonsils or tonsils grade I - II
* Normal finding of larynx and tongue base
* No lingual tonsil hypertrophy
* ASA (American Society of Anaesthesiology, 1963) criteria I or II
* Body mass index (BMI) < 33 kg/m2
* Age > 18 yrs
* Fix bed partner
* Ability to read and understand the patient's information

Exclusion Criteria:

* Previous Pillar implants
* Previous airway surgery other than nasal, adenoid, tonsil or UPPP
* Presence of other sleep disorders
* Psychiatric disorders
* Neurological disorders (e.g. Cerebrovascular injury)
* Dysmorphia of the cranial skeleton
* Pregnancy or breastfeeding
* Known hypersensitivity to nitinol
* Participation in another clinical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2014-04; Primary Completion 2020-07 (Actual); Study Completion 2020-10 (Actual)

PRIMARY OUTCOMES:
Reduction of initial AHI by ≥20% | 90days
  The primary endpoint is the Apnea-Hypopnea-Index (AHI) at the 90 days follow-up.
  Study hypothesis: Reduction of initial AHI ≥20%. AHI is measured using cardio-respiratory polygraphy. Two measurements are performed before treatment and at 90 days follow-up in order to reduce effects from night-to-night variability.

SECONDARY OUTCOMES:
Reduction of initial snoring index ≥30% | 90days
  Endpoint snoring is measured on a continuous Visual Analog Scale (VAS) by the bed partner.
  Study hypothesis: Reduction of initial snoring index ≥30%

CONTACTS AND LOCATIONS:
Overall Officials: Kurt Tschopp, MD, Principal Investigator — Kantonsspital Liestal
Locations (1):
- Kantonsspital Liestal, Basel, Basel-Landschaft, Switzerland